CLINICAL TRIAL: NCT06899581
Title: Monitor Gut Health in Children Undergoing Treatment for Acute Myeloid Leukaemia Treatment: Case-control Study
Brief Title: Gut Health in Children With Cancer
Status: Recruiting | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS345223:23SH27
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: AML (Acute Myelogenous Leukemia; HLH; Burkitt Lymphoma/Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Enteral nutrition Food Derived Ingredient — For this case-control analysis, children with AML will be matched to cancer-free controls for age, sex and race. No antibiotics for 6 months. In collaboration with Professor Konstantinos Gerasimidis Professor of Clinical Nutrition School of Medicine. University of Glasgow. Healthy children have been recruited from the community via poster and social media advertisement. The whole bowel movement was collected in a disposable stool collection kit and stored in a benchtop freezer provided to study participants. Researcher defrosted the sample, homogenised it with mechanical kneading and aliquots were stored in -80.
  Cases: children with AML: Stool specimens will be obtained at three predefined time points for microbiome analysis: baseline start of AML treatment (within 2 weeks of admission); after induction chemotherapy initiation (6-8weeks); recovery phase 6-8 months.

SUMMARY:
The purpose of this study is to observe the impact leukaemia treatment has on gut health (microbiomes) and how quickly the gut health recovers after leukamia treatment. The gut microbiome has a number of important functions not only in the gut but within the whole body. Changes to your child's nutritional status throughout treatment may affect how well they recover from treatment. This study will monitor the impact of feeding and nutrition on nutritional status and gut health in young people undergoing treatment for leukaemia. The measurements needed to observe nutritional and gut microbiomes will occur when your child attends their routine medical appointments at Great Ormond Street Hospital.

Medical treatment uses chemicals to kill leukaemia cells. The type of medications used in the treatment of leukaemia can damage the gut resulting in inflammation call mucositis. This stops the gut from working and sometimes nutrition has to be provided via a feeding tube or intravenous. Chemotherapy, mucositis and intravenous nutrition all have an impact on the gut. Little is know how the gut health recovers after treatment for leukaemia. This will be the first study to specifically monitor the impact of feeding and nutritional on gut health in children undergoing treatment for leukaemia.

By understanding what changes are occurring to your child's nutritional status and gut halth during treatment and during recovery will help to develop guidelines for healthcare professionals to support optimal gut health recovery.

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) is an aggressive cancer that occurs due to the clonal expansion of immature white blood cells, known as blasts (Chaudhury et al., 2018) with generally poor outcomes compared to childhood lymphoid leukaemia (Arad-Cohen et al., 2022). While complete remission rates are high in paediatric AML at approximately 90%, event-free survival and overall survival remain suboptimal at 45% and 65%, respectively, at 3 years, and nearly half of children will relapse (Rasche et al., 2018). Recently there has been a shift towards antigen-targeting immunotherapy in the treatment of cancers, including AML, to trigger anti-leukaemic responses (Greiner, 2019).

Intestinal mucositis is one of the most common side effects of chemotherapy, resulting from disruption of the immunological balance of the intestinal mucosal barrier (De Pietri et al., 2020). This results in alterations of absorptive and secretory functions of the intestinal mucosa, haemorrhages, intestinal dysmotility or intestinal failure (McGrath, 2019; Ohta et al., 2003). Chemotherapy-induced intestinal mucositis is thought to play a central role in the development of systemic inflammation and infections (van der Velden et al., 2014). The clinical assessment of the severity of intestinal mucositis is challenged by the lack of validated scoring scales, and objective biomarkers related to mucositis pathogenesis for assessment of its severity are therefore in demand. Decreasing plasma citrulline levels have been associated with the severity of intestinal mucositis and systemic inflammation after haematopoietic stem-cell transplantation in both adults and children (Gosselin et al., 2014; van Vliet et al., 2009).

Chemotherapy-induced intestinal mucositis causes translocation of intestinal bacteria and allows bacteria to cross the damaged mucosal barrier leading to a systemic inflammation and potentially to systemic infections, especially in immunocompromised patients (Villa and Sonis, 2015). Diseases affecting the immune system, such as inflammatory bowel disease (IBD), juvenile idiopathic arthritis (JIA), and acute leukaemia, are pathological conditions affecting the paediatric population and are often associated with alterations in the intestinal microbiota, such as a decrease in bacterial diversity (Lucafò et al., 2020). Growing evidence suggests that gut microbiota can interfere with chemotherapeutic and immunosuppressant drugs, used in the treatment of these diseases, reducing or facilitating drug efficacy (Peppas et al., 2023). Human intestinal microbiota consists of several hundred bacterial species [(Marchesi et al., 2016)]. The microbial community of the gut conveys significant benefits to human physiology at an intestinal epithelial and systematic inflammatory level [(Kindon et al., 2007; McDonnell et al., 2021) (Feng et al., 2022)].

Feeding strategies in clinical practice in paediatric cancer patients with chemotherapy-induced mucositis varies considerable but invariably requires gut rest and may require parenteral (intravenous) nutrition (Kuiken et al., 2017b)(Kuiken et al., 2017b). Parenteral nutrition is associated with significant adverse effects, namely liver injury, risk of infections, metabolic derangements, gut atrophy, dysbiosis of the intestinal microbiome (Tume et al., 2020) The gut microbiota is the most abundant type of antigen-presenting cells. Therefore, it is conceivable that parenteral nutrition may profoundly alter the gut microbiome composition and function, which could lead to detrimental effects on the intestine (Pierre, 2017).

The catastrophic impact of a fibre-devoid diet on the gut microbial recolonisation post critical illness has been described by Tanes et al,2021, the team outline the importance of introducing the right nutrition after a bout of illness (Tanes et al., 2021). The diversity and relative abundance of microbial metabolites are heavily dependent on specific dietary components [(Morrison and Preston, 2016)]. Non-digestible dietary fiber such as oligosaccharides and inulin demonstrate resistance to digestion in the human small intestine [(Lattimer and Haub, 2010)]. In the large bowel dietary fiber undergoes fermentation by colonic microbiota to produce short chain fatty acids (SCFA); acetate, butyrate and propionate, which act as the primary carbon energy source for colonocyte [5]. The synergistic relationship between the host and intestinal SCFA concentrations include the concomitant reduction of the luminal pH, which by itself inhibits pathogenic microorganisms and increases the absorption of some nutrients [(Macfarlane and Macfarlane, 2012)]. Furthermore, intestinal SCFA control the production of T-helper cells, antibodies, and cytokines and are also involved in maintaining homeostasis of the mucosal system [(Ríos-Covián et al., 2016; Corrêa-Oliveira et al., 2016)].

Dietary and microbiome-based therapies are being explored for the potential to support recovery of healthy gut commensal populations during and after critical illness. In the paediatric population interest is growing in the use of a blended diet for the management of feed intolerances [(Schmitz É et al., 2021)]. Industry have responded to this shift in feeding practices and developed a high fiber enteral formula with food derived ingredients, which has been shown to improve enteral feed tolerance [(O'Connor et al., 2022)].

This is the first study to observe the impact of AML treatment on the gut microbiome of children on different modes of feeding including parenteral nutrition and food-based formulas. Finally, this study will also observe the recovery phase of the gut microbiota after AML treatment and compare with subsequent infections and relapse.

Cases: children with AML: Stool specimens will be obtained at three predefined time points for microbiome analysis: baseline start of AML treatment (within 2 weeks of admission); after induction chemotherapy initiation (6-8weeks); recovery phase 6-8 months.

Paediatric stool samples will be collected using the stool sample collection kit. Each participant will be provided with 4 home collection kits. Each kit contains:

* • Fe-Col® collection kit
* • Stool collection tube (containing stability buffer)
* • Biohazard bag
* • Bubble mailer bag
* • Instructions.

The samples will then be posted back to PeploBio's laboratory (Royal Mail Priority, Track24). Upon arrival, PeploBio personnel will proceed to sample reception, including verification of sample integrity and accessioning. Samples will be homogenized and split into 200ul aliquots and stored for up to 7 days at -20ºC.

Controls: match control stool samples will be sent to PeploBio for microbiome analysis

Assay Summary:

Both case and control stool samples will be sent to PeploBio's Advanced Gut Microbiome Panel offer. This qPCR multiplex assay targets the 16s gene for 10 bacterial targets. These targets will specifically be chosen based on clinical, peer-reviewed correlation studies implicating their involvement in metabolic and inflammatory diseases, such as cancer. The results will provide an absolute quantification data within as little as 1-2 days from sample arrival at the laboratory.

Bioinformatic processing We plan to sequence the V4 region of the bacterial 16S rRNA gene using the Illumina MiSeq platform according to the manufacturer's specifications. Reads will be demultiplexed into fastq files for each sample using sequence barcodes. Forward and reverse reads will be joined with PANDAseq. After samples with fewer than 3000 reads will be excluded. The joined sequence files will be formatted using a Python script to add QIIME headers with the respective sample ID to each sequence before concatenating into one file for input into QIIME 1.8.0A.

The Shannon alpha diversity will be calculated on the unfiltered biom table using the alpha_diversity.py script, and weighted UniFrac distances were calculated with the beta_diversity.py script. The microbial dysbiosis index (initially described by Gevers et al. will be calculated in R for each sample. The microbial dysbiosis index will be defined as the log10 of the total abundance in organisms increased in CD divided by the total abundance of organisms decreased in CD. The increased-in-CD taxa comprise Enterobacteriaceae, Pasteurellaceae, Fusobacteriaceae, Neisseriaceae, Veillonellaceae, and Gemellaceae. Decreased-in-CD taxa are Bacteroidales, Clostridiales (excluding Veillonellaceae), Erysipelotrichaceae, and Bifidobacteriaceae

Gut microbiome composition analysis:

Microbial diversity will be expressed as the number of distinct species in a community (richness), the even distribution of their abundances (evenness) or a combination of both aspects, commonly termed alpha diversity. Microbial alpha diversity is estimated using the Shannon and Simpson indices, whereas microbial richness is estimated using the Chao1 index, or number of observed species/operational taxonomic units (OTUs).

For the extraction of the nucleic acids, the samples are lysed, and nucleic acid extracted using MagMAX™ Viral/Pathogen II (MVP II) Nucleic Acid Isolation Kit, following the manufacturer's IFU (Thermo Scientific). qRT-PCR will be executed using primers designed for the 10 bacterial targets (16s gene), and quantitative absolute abundance is determined using the standard curve method.

Anthropometry (data collection: T0 baseline; T1 end of consolidation 6-8months; T2 Recovery 10-12months) Weight will be determined to the nearest 0.1 kg, with subjects dressed in light clothing or ward gown among patients, using a Model 880 electronic scale (Seca, Hamburg, Germany) after voiding. Height will be measured to the nearest 0.1 cm without socks or shoes, using a Model 206 wall-mounted stadiometer (Seca). Body mass index (BMI) will calculate using the standard formula (kg m-2). Weight and height will be measured following standard procedures. Body mass index will be calculated as weight in kilograms divided by height in meters squared, and BMI SDS will be obtained from the WHO reference curves. BMI and standard deviations scores (SDS) will be calculated using WHO as reference data.

Obesity will be confirmed when the percentile is higher than 99.9th on the WHO Child Growth Standards Curve, or the z-score was higher than +3 (Cole et al., 2000). Children older than 5 years, with BMI between the 85th and 97th percentiles on the WHO Child Growth Standards Curve, will be classified as overweight, and as obese when the percentile is higher than the 97th or the z-score is higher than +2SD. Conversely, underweight will be confirmed when the z-score is lower than -2SD Mid upper arm circumference (MUAC) will be measured halfway between the tip of the acromion and olecranon process using a non-stretchable measuring tape SECA 212 to the nearest 0.1 cm Dietary data collection (data collection: T0 baseline; T1 end of consolidation 6-8months; T2 Recovery 10-12months) Three-day food records will be used to assess dietary intake and enteral nutrition of children. Parents or caregivers will be instructed on how to record the food and fluid consumption of their child using household measures to estimate portion sizes and food type (including brand names of foods, if applicable) in a diary provided. Dietary records will be kept for two weekdays and one weekend day. Analysis of dietary intake will be performed using Nutritics nutritional analysis software (Dublin, Republic of Ireland). Energy and nutrient intake of children will be compared against the SAGN 2017 guidelines (SACN, 2011).

Gastrointestinal Tolerability (data collection: T0 baseline; T1 end of consolidation 6-8months; T2 Recovery 10-12months) Stool consistency is a central component in the description of normal or altered bowel habit. Stool form can be considered as a proxy measure for stool consistency and refers to the shape and apparent texture of the stool, which can be assessed visually. Stool form scales are a standardised and inexpensive method of classifying stool form into a ﬁnite number of categories that can be used by health care professionals and researchers.

Bristol Stool Form Scale is an ordinal scale of stool types ranging from the hardest (Type 1) to the softest (Type 7). Types 1 and 2 are considered to be abnormally hard stools (and in conjunction with other symptoms indicative of constipation) while Types 6 and 7 are considered abnormally loose/liquid stools (and in conjunction with other symptoms indicative of diarrhoea). Type 3, 4 and 5 are therefore generally considered to be the most 'normal' stool form and are the modal stool forms in cross-sectional surveys of healthy adults. [22] Tolerance and details of stooling patterns will be recorded each week at a ward level and at home depending on treatment phase. Descriptions of feeding intolerance will include a report of the following variables: stool consistency and volume (number of stools in a 24-hour period), abdominal distension, gas, vomiting, and overall comfort level of the patient.

Other sources of data collection:

Impact of Chemotherapy

* Length of intestinal mucositis
* Length of time of parenteral (intravenous) nutrition
* Length of time on enteral nutrition including nutritional composition of formula
* Infection and antibiotic use
* Any other significant medical event related to treatment

STUDY SETTING Single centre tertiary haematology centre - Great Ormond Street Hospital. Sampling

Data analysis strategies Sample size calculated on primary outcome - alpha diversity primary outcome marker: The sample size calculations will be based on the association between total microbial alpha-diversity (the richness and evenness) to find the difference in diversity between control and case participants post-treatment for AML (end of induction - 1 month) Assuming an adequate power (80%), a total of 50 samples (25 per group) will be required for an effect size of 0.82.

(Mattiello et al., 2016). Microbial Diversity in Clinical Microbiome Studies: Sample Size and Statistical Power Considerations (gastrojournal.org)

25 children control (1 stool samples) 25 children cases (3 timepoints = 75 stool samples)

Alpha diversity associations with case-control status will be tested by linear and unconditional logistic regression, with adjustment for age and sex. Composition of the microbiota (beta diversity) will be compared by unweighted and weighted UniFrac analysis of the distance matrix with 10 000 permutations. The Mann-Whitney U test will be used for comparisons of diversity and ratios of component bacteria at the genus and species levels. Relative abundance of the microbes will be expressed as median ± range and a Wilcoxon signed-rank test will be used for comparison of alpha diversity in case vs. control at baseline and 6 months follow-up and comparison of relative abundance between baseline and later time points.(Plaza-Díaz et al., 2019).

The Wilcoxon rank sum test was used for comparison between groups, whereas permutational multivariate analysis of variance (PERMANOVA) was used to evaluate the gut microbiota composition at the OTU and genus level.

Changes in Microbiota Diversity and Composition During Chemotherapy: A linear mixed-effects model examined changes in the diversity indices using R version 4.3.1. For microbiome compositional change, a mixed-effects negative binomial regression model will be used The P value will be adjusted for the false discovery rate with the Benjamini-Hochberg method and reported as Q value (Benjamini and Hochberg, 1995).

Normality will be checked using the Shapiro-Wilk test in the coin-package of R (Hothorn et al., 2006). The non-parametric multivariate analyses of variance tests will be performed by Adonis function which will be set to 9999 permutations. Data will be summarized according to their respective distribution. For parametric data, means ± SD (standard deviation), for non-parametric variables, medians ± IQR (inter-quartile range) are presented. For all statistical analyses, the significance level will be based on P-value ≤ 0.05.

Impact of Baseline Microbiota on Infection Outcomes For initial risk stratification at the time of AML diagnosis, the Wilcoxon-Mann-Whitney test and logistic regression will be used to assess potential risk factors for subsequent infection occurring at any time during the study period, including the baseline microbiome. For each taxon whose relative abundance significantly differed among patients who had or did not have the event, the RA will be dichotomized at the optimal cutoff value based on the Youden index. Factors with a P value of <.1 in univariate analysis will be examined by multiple logistic regression. The cumulative incidence of outcomes will be compared among risk factors with Gray test.

7.3 Recruitment The researchers will attend ward rounds and view EPIC (electronic notes) each day to identify new admission with ALL Families will be identified at ward level by their dietitian a member of the patient's existing clinical care team who will check whether they meet the inclusion criteria in light of requiring enteral tube feeding for children who display signs of feed intolerance. An initial approach with a letter of invitation and a participant information sheet will be given to them explaining the study with the details of the research team to discuss the feeding options on the study 7.3.1 Sample identification Consent The study's participant information sheet will be offered to the potential participant's family member/carer accompanied by an age-appropriate information sheet describing: the study; its purpose and nature, what it will require for the participant; its risks and burdens, the propositions and limitations of the protocol; the known side effects and any risks involved in taking part. It will be clearly stated that participation is entirely voluntary, be able to make a free choice and the participant is free to withdraw from the study at any time for any reason without affecting or impacting their care, without affecting their rights, and with no requirement to justify withdrawal. This is clearly outlined in the opening paragraphs of PIS.

The participant will be allowed 3 days to consider the information, and the chance to ask any question to the Investigator. Written Informed Consent from the participant's representative will be required and then obtained and the person obtaining the consent must be appropriately qualified, experienced and authorised to do so by the Chief/Principal Investigator.

Informed Consent/Assent Process A signed copy of the study informed consent /assent form will be given to the participant's legal representative and a copy in the participant's medical records. An original signed form will be retained at the study site in a secure place. Competent Adults (aged 16 at the time of consent) Upon completion of the above, the patient will then sign and date the informed consent document. Both the person obtaining consent and the participant must personally sign and date the form. A copy of the informed consent document will be given to the patient for their records. The original copy will be filed in the participant's medical notes and a further copy of the signed consent form will be filed in the Investigator Site File. One copy of the consent form should be sent to the YP (aged <16 years at the time of consent) informed consent for a young person under the age of 16 years is provided by a person with parental responsibility or a legal representative.

Children aged 6 years and above will be approached for assent unless the clinical care team deem otherwise, then they will not be entered into the study until assent (in addition to legal consent from an appropriate adult) is provided - an exception to this is made where the minor expresses a wish for the decision to be made solely by the appropriate adult.

Age-appropriate REC-reviewed information Sheets and assent forms, that have been given a favourable opinion, describing (in simplified terms) the details of the study intervention, study procedures and risks will be available for use. The YP should personally write their name and date on the assent form, which is then signed by the parent/legal representative and the researcher.

Young people who were under 16 years old when treatment initially started and turn 16 years old while on the study will be re-consented using specific PIS and consent forms Consent (hard copies) forms will be uploaded into the electronic notes (EPIC) and hard copy stored in the dietetics office in a locked draw during the study. Once the study is closed, consent forms will be transferred to the R&D Achieves Dietetic Research Storage - £25 annual fee covered by dietetics.

Participants who may have difficulties in an adequate understanding of English will be supported by GOSH Trust interpretation service. 'Thebigword' is the Trust's sole supplier of telephone interpreting, a service which will enable you to help any client who may have limited English language skills. 0800 694 5093 The consent will be recorded in a patient's electronic notes and in the study records.

8 ETHICAL AND REGULATORY CONSIDERATIONS This protocol and related documents will be submitted for ethics review to Integrated Research Application System (IRAS) and Health Research Authority (HRA).

Assessment and management of risk

8.1 Research Ethics Committee (REC) and other Regulatory review & reports

* Before the start of the study, a favourable opinion will be sought from a REC
* Before the start of the study, approval from the Health Research Authority (HRA) and Health and Care Research Wales (HCRW) for project-based research taking place in the NHS in England and Wales will be sought.

For NHS REC reviewed research

* Substantial amendments that require review by NHS REC and HRA will not be implemented until that review is in place and other mechanisms are in place to implement at site.
* All correspondence with the REC and HRA will be retained.
* It is the Chief Investigator's responsibility to produce the annual reports as required.
* The Chief Investigator will notify the REC of the end of the study.
* An annual progress report (APR) will be submitted to the REC within 30 days of the anniversary date on which the favourable opinion was given, and annually until the study is declared ended.
* If the study is ended prematurely, the Chief Investigator will notify the REC, including the reasons for the premature termination.
* Within one year after the end of the study, the Chief Investigator will submit a final report with the results, including any publications/abstracts, to the REC.

Regulatory Review & Compliance

* This is a single-centre study
* Before any site[s] can enrol patients into the study, the Chief Investigator/Principal Investigator or designee will ensure that appropriate approvals from participating organisations are in place.
* For any amendment to the study, the Chief Investigator or designee, in agreement with the sponsor will submit information to the appropriate body in order for them to issue approval for the amendment. The Chief Investigator or designee will work with sites (R&D departments at NHS sites as well as the study delivery team) so they can put the necessary arrangements in place to implement the amendment to confirm their support for the study as amended.

ELIGIBILITY:
Inclusion Criteria:

* - Consented to partake in the study
* Aged 0-16 years old
* Diagnosed with AML/HLH/ Burkits

Exclusion Criteria:

* 17 years old + (treated at UCL adolescent unit)
* Inflammatory bowel disease: ulcerative colitis or Crohn's disease
* Children who had previously been treated with chemotherapy in another institution age

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | 6 months
  (1a) differences in the alpha and beta-diversity throughout AML treatment and recovery phases
  1. b) differences in the alpha and beta diversity at baseline between case and controls
  2. a) differences in the Firmicutes to Bacteroidetes ratio throughout AML treatment and recovery phases
  (2b) differences in the Firmicutes to Bacteroidetes ratio baseline between case and controls (3a) differences in gut microbiome composition throughout AML treatment and recovery phases (3b) differences in gut microbiome composition baseline between case and controls

SECONDARY OUTCOMES:
Anthropometry | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Nov 2026